CLINICAL TRIAL: NCT03941847
Title: Musinduc : Impact of Music During the Period of Anaesthetic Induction - a Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Musical Listening on Hypnotic Savings During the Induction of General Anesthesia
Acronym: MUSINDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHU 19-007
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2020-01

CONDITIONS: Music, Anesthetic, Induction
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups will be compared. The experimental group will benefit from musical listening during the induction period of the anesthesia. The control group will have a usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- music (Experimental): The experimental group will benefit from musical listening during a classic period of induction of anesthesia
  Interventions: Other: music
- silence (No Intervention): The control group will have a usual care.

INTERVENTIONS:
Other: music — listening music
  Arms: music

SUMMARY:
Anesthetic induction requires the use of, among other things, hypnotic drugs that can lead to hemodynamic disorders, postoperative cognitive dysfunctions and delayed awakening. A strategy to reduce the doses of hypnotics administered could improve patients' postoperative outcomes and is part of the current strategy of accelerated postoperative rehabilitation. Music has shown its effectiveness in reducing the doses of hypnotics administered during sedation procedures.

Objective :

We propose a study of this anesthetic period evaluating the effectiveness of music as an adjuvant agent for anesthetic drugs allowing hypnotic savings.

Materials and methods :

Randomized, prospective, monocentric study

2 groups will be compared. The experimental group will benefit from musical listening during the induction period of the anesthesia. The control group will have a usual care.

The primary endpoint is the amount of hypnotic (propofol®) used during anesthesia induction. The main secondary criteria are the duration of induction, the cost of induction, and the postoperative pain score and the proportion of patients with postoperative nausea and vomiting.

This study should include 104 subjects (52 in each group) requiring general anesthesia.

Hypothesis tested:

Listening to music reduces the amount of hypnotic product used in the induction of anesthesia by 0.5 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for surgery under general anesthesia in ophthalmic surgery, ENT, CMF and neurosurgery (lumbar and cervical disc hernia, neurostimulator insertion, vertebral cementoplasty)
* Score ASA 1, 2, 3.
* Intervention time < 3 hours.

Exclusion Criteria:

* Patients under 18 years of age
* Patient under guardianship or curatorship
* Refusal of the patient
* Deaf patient
* Non-cooperating patient
* Anesthetic protocol different from that standardised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
quantity of propofol | 2 months
  quantity of propofol in mg/kg necessary for the induction of general anaesthesia

SECONDARY OUTCOMES:
Quantity of morphinomimetics | 2 months
  Quantity of morphinomimetics (morphine equivalent) used in mg for anesthetic induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Uteza, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No